CLINICAL TRIAL: NCT05422456
Title: The Turkish Adaptation, Validity, and Reliability of the Functional Disability Inventory
Brief Title: The Turkish Version of Functional Disability Inventory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2022-126
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: pediatric; chronic pain; headache; functional disability
MeSH Terms: conditions — Chronic Pain; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pain group: children are diagnosed with chronic headache by pediatric neurologist
- Health group: children without chronic pain

SUMMARY:
The goal of this study is to determine the validity and reliability of the Turkish version of the Functional Disability Inventory (FDI), which assesses functional disability in daily life, school, and home activities of children aged 8 to 18, as well as to ensure cultural adaptation of this measurement. Chronic pain is the most frequent type of pain in children and adolescents, affecting one-quarter of the population. Children and adolescents with chronic pain have difficulty completing activities such as walking, jogging, and participating in sports, as well as daily activities. There is no valid and reliable measurement that measures pain-related disability in everyday life, at home, or at school from the perspective of a child in the literature. This study hypothesizes that the Functional Disability Inventory is a valid and reliable measurement for measuring functional disability in the Turkish population of children with chronic pain.

DETAILED DESCRIPTION:
Chronic pain in children and adolescents is defined as pain that lasts longer than three months and is unabsorbable. Approximately 5% of the children said they were suffering from moderate to severe chronic pain, as well as impairments in their physical and psychosocial functions. Children and adolescents with chronic pain have difficulty completing activities such as walking, jogging, and participating in sports, as well as daily activities. Schoolchildren with chronic pain, for example, were shown to be five times more likely than their classmates without pain to miss school (13.9 percent vs. 2.4 percent), and it has been observed that absenteeism from school increases the likelihood of grade repeat in children with chronic pain.

Headaches affect between 57 and 82 percent of children and adolescents aged 7 to 15. It is wrong to believe that a headache with this frequency and associated concomitant conditions does not result in functional disability and limitations in everyday activities. When compared to their peers without headaches, 62 percent of children and adolescents with headaches reported more functional disability due to moderate to severe headache, limitation in daily activities, and absenteeism from school. Pain and functional incapacity caused by pain cannot be assumed to have no impact on a person's ability to participate in activities. The term "participation" refers to a person's involvement in the circumstances of his or her life. Participation in daily activities is critical for all children's healthy development, regardless of their age.

The fundamental goal of functional evaluation is to demonstrate a person's ability to function in society independently. This skill is employed in everyday activities such as personal care, social contact, housework, and recreational activities. The importance of these functions in daily life in pediatric patients, on the other hand, receives less emphasis (5). Walker and Greene (1991) developed the Functional Disability Inventory (FDI) to assess impairments in children and adolescents caused by a variety of pediatric health conditions (6). There are fifteen items in the FDI category. These tasks are used to assess how difficult it is for the youngster to walk, climb stairs, eat, do household chores, go to school, participate in sports, read and write, and watch television.

On a four-point Likert scale, (0=no issue, 4=impossible), each item is rated. With the child's own report, FDI assesses the difficulty in physical and psychological functions caused by the child's physical health. It is determined by taking into account the child's activity restrictions throughout the previous two weeks. The scale runs from 0 to 60. The total score is calculated by summing the individual item scores. A higher score indicates a higher level of disability. The purpose of this study is to see if the Turkish version of the Functional Disability Inventory (FDI) is valid and reliable in a Turkish sample of children with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pain
* Age between 8-18 years
* Native language is Turkish

Exclusion Criteria:

- Diagnosis of autism spectrum disorder and attention deficit and hyperactivity disorder, psychotic symptoms, depression, etc.

Inclusion Criteria for control group:

* Not diagnosed of chronic pain and psychiatric and neurological disease
* Aged at 8-18 years old
* Native language is Turkish

Exclusion Criteria for control group:

* Children whose parents or themselves refused to participate
* Native language is not Turkish

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children are diagnosed with chronic headache and their health peers
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional disability | Baseline
  Functional Disability Inventory (FDI) is 15 item self-report measurement designed to evaluate functional disability in children while they were doing various activities. Each item scored 0 to 4; 0 represents no trouble and 4 represents impossible.
Evaluation of severity of pain | Baseline
  Wong-Baker Face Pain Scale is valid and reliable measurement preferred by children and parents to evaluate severity of pain. It consists of 6 face expression that symbolized pain severity. These Show the stages of increased pain from smiling face (0 point) to a very sad and crying face (10 points). Children rate their current pain between these faces.
Evaluation of pain | Baseline
  In several pediatric diagnostic groups, the Adolescent Pediatric Pain Tool (APPT) is applied for pain assessment APPT can be used on children aged 7 to 18. The APPT consists of three separate parts. First, the body diagram allows the child to indicate the location of the pain. Second, pain intensity was rated on a scale from "no pain" to "worst possible pain" based on 5-point Likert scale. Finally, the characteristics of pain and 67 words describing pain are indicated.

SECONDARY OUTCOMES:
Evaluation of somatization | Baseline
  Children's Somatization Inventory is a scale that evaluates the child's symptoms experienced in the last two weeks in both parent and child forms and the child's somatization symptoms from both perspectives. Total score is obtained by adding up all the scores. Higher scores indicate greater somatization complaints. Scores range from 0 to 96.
Evaluation of quality of life | Baseline
  Pediatric Quality of Life Inventory is a generic health related quality of life measure consisting of four core scales, physical function (8 items), emotional function (5 items), social function (5 items) and school function (5 items) that is intended for use in healthy and patient populations. Respondents are asked to recall the last month and indicate how frequently - from never to almost always - they have experienced specific phenomena. Item responses (0-100) are averaged to form total and core scores; higher scores indicate higher functioning.
Evaluation of anxiety | Baseline
  The measurement consists of two subscales as State Anxiety Scale and Trait Anxiety Scale. Each subscale has 20 items, and 40 items in total. State Anxiety scale assesses momentary subjective feelings in certain situations. Trait Anxiety Scale assesses continued subjective chronic feelings such as worry, anxiety and irritability. Total scores change between 20-80. Scores between 20-39 indicate mild, scores between 40-59 indicate moderate, scores between 60-79 indicate severe anxiety, and scores of 80 indicate panic.
Evaluation of Depression | Baseline
  Children Depression Scale is a measurement that can be used in children aged 6-17. The scale evaluates using the child's own answers. It consists of 27 items. In these choices, there are "sometimes," "often" and "always" answers containing the item related to the question. Each item scored with 0,1,2. The highest score is 54, and higher scores indicating higher level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the results will be published in the journal

REFERENCES:
- [Result] Murphy NA, Carbone PS; American Academy of Pediatrics Council on Children With Disabilities. Promoting the participation of children with disabilities in sports, recreation, and physical activities. Pediatrics. 2008 May;121(5):1057-61. doi: 10.1542/peds.2008-0566. PMID 18450913
- [Result] Sonagra M, Jones J, McGill M, Gmuca S. Exploring the intersection of adverse childhood experiences, pediatric chronic pain, and rheumatic disease. Pediatr Rheumatol Online J. 2022 Feb 14;20(1):14. doi: 10.1186/s12969-022-00674-x. PMID 35164793
- [Result] Offenbacher M, Kohls N, Walker L, Hermann C, Hugle B, Jager N, Richter M, Haas JP. Functional limitations in children and adolescents suffering from chronic pain: validation and psychometric properties of the German Functional Disability Inventory (FDI-G). Rheumatol Int. 2016 Oct;36(10):1439-48. doi: 10.1007/s00296-016-3504-5. Epub 2016 Jun 4. PMID 27262712
- [Result] Groenewald CB, Tham SW, Palermo TM. Impaired School Functioning in Children With Chronic Pain: A National Perspective. Clin J Pain. 2020 Sep;36(9):693-699. doi: 10.1097/AJP.0000000000000850. PMID 32487871
- [Result] Ferracini GN, Dach F, Speciali JG. Quality of life and health-related disability in children with migraine. Headache. 2014 Feb;54(2):325-34. doi: 10.1111/head.12251. Epub 2013 Oct 29. PMID 24512577
- [Result] Claar RL, Walker LS. Functional assessment of pediatric pain patients: psychometric properties of the functional disability inventory. Pain. 2006 Mar;121(1-2):77-84. doi: 10.1016/j.pain.2005.12.002. Epub 2006 Feb 9. PMID 16480823
- [Derived] Koklukaya HN, Kaya Kara O, Karademir S, Dogan M, Kutluk MG, Kara K. An evaluation of the validity, reliability, and psychometric properties of the Turkish version of the functional disability inventory in children and adolescents with chronic pain. J Pediatr Nurs. 2025 May-Jun;82:e126-e133. doi: 10.1016/j.pedn.2025.04.005. Epub 2025 Apr 17. PMID 40251104